CLINICAL TRIAL: NCT04908761
Title: Quadratus Lumborum Block for Analgesia After Living Donor Kidney Transplantation: A Randomized Controlled Trial
Brief Title: Quadratus Lumborum Block After Living Donor Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun-Kyung Park, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2104-083-1211
Record Dates: First submitted 2021-05-20; First posted 2021-06-01 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Single center, double-blind, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, medical staff who measure outcome variables, and nurses in the recovery room are double-blinded so that medical staff and patients do not know the patient's assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transmuscular quadratus lumborum block group (Experimental): Patients assigned to the Transmuscular Quadratus Lumborum (TQL) block group receive the Transmuscular Quadratus Lumborum block in a lateral decubitus position with the surgical site facing up before recovery of general anesthesia after surgery. For the block, 30cc of 0.375% ropivacaine is used.
  Interventions: Procedure: Transmuscular quadratus lumborum block
- Control group (Placebo Comparator): For patients assigned to the control group, 30cc of 0.9% normal saline is used for Transmuscular Quadratus Lumborum block.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Transmuscular quadratus lumborum block — Patients assigned to the TQL block group receive the TQL block in a supine position with the surgical site facing up before recovery of general anesthesia after surgery. For the block, 30cc of 0.375% ropivacaine is used.
  Arms: Transmuscular quadratus lumborum block group
Procedure: Placebo — For patients assigned to the control group, 30cc of 0.9% normal saline is used for TQL block.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the postoperative analgesic effect of quadratus lumborum block in patient undergoing a living donor kidney transplant under general anesthesia.

DETAILED DESCRIPTION:
The purpose of this study was to investigate whether postoperative pain is significantly reduced when TQL block was additionally performed after surgery in patients undergoing living-donor kidney transplantation. Therefore, investigator hypothesized that the analgesic consumption for postoperative 24 hours will decrease in TQL group compared to the control group. For secondary outcomes, the pain score at rest/ movement up to 48 hours after surgery, the time until the first pain reliever is requested, whether and how often rescue analgesics are administered for 48 hours, the incidence and severity of nausea and vomiting during the 48 hours after surgery, patient's satisfaction with post-pain control and the number of hospital stays were investigated. Overall, the aim of this study is to evaluate the postoperative analgesic effect of quadratus lumborum block in patients undergoing a living donor kidney transplantation under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years of age undergoing elective living donor kidney transplantation under general anesthesia in Seoul National University Hospital

Exclusion Criteria:

* Patients with severe pain before surgery

  * Patients with a history hypersensitivity reactions on fentanyl or ropivacaine

    * Patients who cannot maintain patient-controlled analgesia (PCA) by themselves

      ④ Patients with skin diseases or infections in the area where quadratus lumborum block is applied

      ⑤ Any other cases that researchers determine that it is inappropriate for this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption for 24 postoperative hours | 24 hours postoperatively
  Total analgesic use for 24 hours after surgery (morphine milligram equivalents (MME))

SECONDARY OUTCOMES:
Analgesic consumption | at postoperative 6, 12, 48 hours
  Analgesic consumption at postoperative 6, 12, 48 hours
Resting pain numeric rating scale(NRS) | at postoperative 6, 12, 24, 48 hours
  Resting pain numeric rating scale(NRS) at postoperative 6, 12, 24, 48 hours. Numeric rating scare is 11-point scale from 0 to 10, The higher the number, the more severe the pain (0 is no pain at all, 10 is the most severe pain imaginable).
Numeric rating scale of pain during movement | at postoperative 6, 12, 24, 48 hours
  Numeric rating scale of pain during movement at postoperative 6, 12, 24, 48 hours Numeric rating scare is 11-point scale from 0 to 10. The higher the number, the more severe the pain (0 is no pain at all, 10 is the most severe pain imaginable).
Time to first rescue analgesics | within post-operative 24 hours
  Time to first rescue analgesics
Numeric rating scale at post anesthetic care unit (PACU) | 30 minutes after the end of operation
  Numeric rating scale at post anesthetic care unit Numeric rating scare is 11-point scale from 0 to 10. The higher the number, the more severe the pain (0 is no pain at all, 10 is the most severe pain imaginable).
Rescue analgesics administration | within post-operative 48 hours
  Rescue analgesics administration count
The incidence of post-operative nausea and vomiting | within post-operative 48 hours
  The incidence of post-operative nausea and vomiting
Patient satisfaction with pain control | At post-operative 48 hours
  Patient satisfaction with pain control in 11 point scale (0-10), The higher the score, the higher the patient's satisfaction.
Pattern of injectate spread on ultrasonography | During procedure quadratus lumborum (QL) block
  Pattern of injectate spread on ultrasonography
Sensory blockade | 30 minutes after the end of operation
  After surgery, an alcohol swab is used to evaluate the loss of cold sensation. It is evaluated by dividing into nine regions bordering the rib margin on the side of the surgery, the horizontal line passing through the umbilicus and pubis, and the vertical line of the midclavicular line, anterior axillary line, and mid axillary line. If cold sensation is the same as the opposite part of the regions, marked as 2 points, if decreased marked as 1 point, and if not sensed at all, marked as 0 point.
Quality of Recovery Questionnaire (15-item Quality of Recovery) | At post-operative 48 hours
  Each item uses an 11-point numeric rating scale. The sum of the scores of the 15 items ranges from 0 to 150, with a high score indicating good quality of recovery.
The severity of post-operative nausea and vomiting | within post-operative 48 hours
  The severity of post-operative nausea and vomiting, The severity of the nausea and vomitting is asked to patient and expressed as none, mild, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Kyung Park, M.D.,Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang P, Luo Y, Lin L, Zhang H, Liu Y, Li Y. The efficacy of transversus abdominis plane block with or without dexmedetomidine for postoperative analgesia in renal transplantation. A randomized controlled trial. Int J Surg. 2020 Jul;79:196-201. doi: 10.1016/j.ijsu.2020.05.073. Epub 2020 Jun 2. PMID 32502705
- [Background] Territo A, Mottrie A, Abaza R, Rogers C, Menon M, Bhandari M, Ahlawat R, Breda A. Robotic kidney transplantation: current status and future perspectives. Minerva Urol Nefrol. 2017 Feb;69(1):5-13. doi: 10.23736/S0393-2249.16.02856-3. Epub 2016 Nov 30. PMID 28009142
- [Background] Kruszyna T, Niekowal B, Krasnicka M, Sadowski J. Enhanced Recovery After Kidney Transplantation Surgery. Transplant Proc. 2016 Jun;48(5):1461-5. doi: 10.1016/j.transproceed.2015.11.037. PMID 27496428
- [Background] Freir NM, Murphy C, Mugawar M, Linnane A, Cunningham AJ. Transversus abdominis plane block for analgesia in renal transplantation: a randomized controlled trial. Anesth Analg. 2012 Oct;115(4):953-7. doi: 10.1213/ANE.0b013e3182642117. Epub 2012 Jul 4. PMID 22763899
- [Background] Rohan VS, Taber DJ, Patel N, Perez C, Pilch N, Parks S, Bolin E, Nadig SN, Baliga PK, Fleming JN. Impact of a multidisciplinary multimodal opioid minimization initiative in kidney transplant recipients. Clin Transplant. 2020 Oct;34(10):e14006. doi: 10.1111/ctr.14006. Epub 2020 Sep 4. PMID 32524643
- [Background] de Boer HD, Detriche O, Forget P. Opioid-related side effects: Postoperative ileus, urinary retention, nausea and vomiting, and shivering. A review of the literature. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):499-504. doi: 10.1016/j.bpa.2017.07.002. Epub 2017 Jul 8. PMID 29739538
- [Background] Jun JH, Kim GS, Lee JJ, Ko JS, Kim SJ, Jeon PH. Comparison of intrathecal morphine and surgical-site infusion of ropivacaine as adjuncts to intravenous patient-controlled analgesia in living-donor kidney transplant recipients. Singapore Med J. 2017 Nov;58(11):666-673. doi: 10.11622/smedj.2017077. Epub 2017 Aug 14. PMID 28805236
- [Background] Korgvee A, Junttila E, Koskinen H, Huhtala H, Kalliomaki ML. Ultrasound-guided quadratus lumborum block for postoperative analgesia: A systematic review and meta-analysis. Eur J Anaesthesiol. 2021 Feb 1;38(2):115-129. doi: 10.1097/EJA.0000000000001368. PMID 33186305
- [Background] Uppal V, Retter S, Kehoe E, McKeen DM. Quadratus lumborum block for postoperative analgesia: a systematic review and meta-analysis. Can J Anaesth. 2020 Nov;67(11):1557-1575. doi: 10.1007/s12630-020-01793-3. Epub 2020 Aug 17. PMID 32808097
- [Derived] Kim Y, Kim JT, Yang SM, Kim WH, Han A, Ha J, Min S, Park SK. Anterior quadratus lumborum block for analgesia after living-donor renal transplantation: a double-blinded randomized controlled trial. Reg Anesth Pain Med. 2024 Aug 5;49(8):550-557. doi: 10.1136/rapm-2023-104788. PMID 37704438